CLINICAL TRIAL: NCT00200161
Title: A Randomized Phase II Trial of Concurrent Temozolomide and Radiotherapy Followed by Dose Dense Versus Metronomic Temozolomide and Maintenance Cis-Retinoic Acid for Patients With Newly Diagnosed Glioblastoma and Other Malignant Gliomas
Brief Title: Temozolomide & RT Followed by Dose Dense vs Temozolomide & Retinoic Acid in Pts w/Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Schering-Plough (Industry); Columbia University (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-079
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2016-09

CONDITIONS: Glioblastoma; Gliomas
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Temozolomide

ARMS (2):
- Metronomic Therapy Cohort (Active Comparator): Concurrent temozolomide and radiotherapy plus lose dose of temozolomide
  Interventions: Drug: Temozolomide
- Dose-Dense Therapy Cohort (Experimental): Concurrent temozolomide and radiotherapy plus high dose of temozolomide
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Focal RT 6000 cGy/ Temozolomide 75 mg/m2 then Temozolomide 50mg/m2 will be given to patients on days 1-28 of each 28 day cycle. Maintenance cis-retinoic acid. This therapy will start at the completion of 6 cycles of adjuvant temozolomide in all patients who have had no clinical or radiographic evidence of tumor progression.Treatment will continue in 28 day cycles until tumor progression.
  Arms: Metronomic Therapy Cohort
Drug: Temozolomide — Focal RT 6000 cGy/ Temozolomide 75 mg/m2 plus Temozolomide 150 mg/m2 will be given to patients on days 1-7 and 15-21 of each 28 day cycle. Maintenance cis-retinoic acid. This therapy will start at the completion of 6 cycles of adjuvant temozolomide in all patients who have had no clinical or radiographic evidence of tumor progression.Treatment will continue in 28 day cycles until tumor progression.
  Arms: Dose-Dense Therapy Cohort

SUMMARY:
Patients have a newly diagnosed brain tumor called a malignant glioma and participate in the study to see if it is possible to increase the benefit of temozolomide when given after radiation. A recent study showed that patients with newly diagnosed glioblastoma lived longer when treated with both temozolomide and radiotherapy followed by 6 months of temozolomide than patients treated with radiotherapy alone. Patients will receive standard low dose temozolomide during radiation. After radiation, they will be randomized to receive either more intense temozolomide or continuous low dose temozolomide.

DETAILED DESCRIPTION:
This is a randomized phase II study that will test two different adjuvant temozolomide regimens in patients with newly diagnosed glioblastoma multiforme. The goal of this study is to identify a regimen that would be appropriate to bring to a phase III trial and compare to the standard dosing regimen of temozolomide recently reported by Stupp et al. in the New England Journal of Medicine. Secondary goals of this study include: prospective analysis of the prognostic impact of MGMT status and generation of preliminary data regarding this treatment strategy for other types of malignant glioma.

The decision regarding which treatment patients receive is made randomly. Neither them or their doctor can select which treatment the patient will receive. There is reason to believe that both of these doses may benefit treating your brain tumor. After 6 months of chemotherapy, and assuming the brain tumor has not shown any sign of growth, they will begin receiving cis-retinoic acid. Cis retinoic acid has been shown in one study to possibly prevent or delay tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of a malignant glioma.
* Tissue block or unstained slides must be available for MGMT analysis.
* Age 18-70
* KPS > 50
* Granulocyte count >1.5 X 109/L
* Platelet count >99 X 109/L
* SGOT < 2.5X upper limit of normal (ULN).
* Serum creatinine < 2X ULN.
* Bilirubin < 2X ULN.
* All patients must sign written informed consent.

Exclusion Criteria:

* Any prior chemotherapy, radiotherapy and biologic therapy for glioma.
* Any prior experimental therapy for glioma.
* Other concurrent active malignancy (with the exception of cervical carcinoma in situ or basal cell ca of the skin).
* Serious medical or psychiatric illness that would in the opinion of the investigator would interfere with the prescribed treatment.
* Pregnant or breast feeding women.
* Refusal to use effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2005-08-09; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa DeAngelis, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 85 participants had a Glioblastoma diagnosis.
  The remaining participants consist of an exploratory cohort of Grade 3 tumors.
Period: Overall Study
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort
Started | 43 | 42
Completed | 43 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Median (Full Range); unit: years] | 54.1 [21 to 71] | 59.1 [30 to 70] | 56.3 [21 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 40 | 82
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 37 | 37 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Overall Survival of Patients With Newly Diagnosed Glioblastoma Multiforme Treated With Concurrent Temozolomide and Radiotherapy Followed by Dose Dense or Metronomic Dosing of Temozolomide and Maintenance Cis-retinoic Acid.
Time Frame: until death or date of last follow up, an average of 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort
Number analyzed (Participants) | 43 | 42
percentage of participants | 69 | 80

2. Secondary Outcome: Progression Free Survival at 6 Months
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort
Number analyzed (Participants) | 43 | 42
percentage of participants | 46 | 56

3. Secondary Outcome: Prognostic Impact of Methylated MGMT Status.
Description: MGMT promoter methylation is currently considered the main prognostic biomarker in glioblastoma. Methylation MGMT status will be assessed using real-time PCR.
Time Frame: through study completion, an average of 1 year
Population: Data were not collected
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: To Collect Preliminary Data on the Efficacy of This Regimen and Impact of MGMT Status in Other Malignant Glioma Subtypes.
Time Frame: through study completion, an average of 1 year
Population: Data were not collected
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Metronomic Therapy Cohort | Dose-Dense Therapy Cohort
All-Cause Mortality (participants affected / at risk) | 0/43 | 1/42
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 43/43 | 42/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metronomic Therapy Cohort (N=43) | Dose-Dense Therapy Cohort (N=42)
Bilirubin (Investigations) | 22 | 18
Hyperglycemia (Metabolism and nutrition disorders) | 34 | 32
Alkaline Phosphatase (Investigations) | 10 | 8
ALT (Investigations) | 43 | 36
Lymphopenia (Investigations) | 30 | 27
PTT (Investigations) | 7 | 8
Muscle weakness - right sided (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness - Left sided (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness extremity - lower (Musculoskeletal and connective tissue disorders) | 0 | 2
AST (Investigations) | 24 | 14
Platelets (Investigations) | 35 | 27
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 | 26
Thrombosis (Vascular disorders) | 8 | 1
Hyponatremia (Metabolism and nutrition disorders) | 13 | 15
Hemoglobin (Blood and lymphatic system disorders) | 33 | 23
Hypokalemia (Metabolism and nutrition disorders) | 12 | 12
Creatinine (Investigations) | 6 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatremia (Metabolism and nutrition disorders) | 15 | 14
INR (Investigations) | 7 | 11
Seizure (Nervous system disorders) | 4 | 4
Constipation (Gastrointestinal disorders) | 5 | 5
Headache (Nervous system disorders) | 7 | 6
Urinary Frequency (Renal and urinary disorders) | 2 | 2
Leukocytes (Blood and lymphatic system disorders) | 16 | 24
ANC (Investigations) | 9 | 13
Hypomagnesmia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 | 3
Amylase (Investigations) | 3 | 1
Lipase (Investigations) | 4 | 0
Infection (Infections and infestations) | 2 | 1
Edema: limb (General disorders) | 0 | 2
Fatigue (General disorders) | 11 | 20
Tremor (Nervous system disorders) | 2 | 0
Fatigue (General disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 3
Hypercholesterolemia (Investigations) | 6 | 5
Speech impairment (Nervous system disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Depression (Psychiatric disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Blurred vision (Eye disorders) | 1 | 4
Confusion (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT00200161/Prot_SAP_000.pdf